CLINICAL TRIAL: NCT00247819
Title: Allelic Linkage in Substance Abuse
Brief Title: The Genetic Basis for Vulnerability to Substance Abuse
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: NIDA-IRP-148
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-10

CONDITIONS: Substance Abuse
Keywords: Substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood draw

SUMMARY:
This investigation seeks to better define the genetic basis for vulnerability to substance abuse.

DETAILED DESCRIPTION:
Dopamine (DA), a neurotransmitter helping to mediate reward and reinforcement, has been putatively linked to the development of substance abuse, alcohol abuse, and alcoholism. Identification of specific vulnerability-association alleles for receptors, other molecules within the reward mediating system, and other genes that may predispose individuals to the development of such disorders is the goal of the study.

This investigation will help elucidate the genetic underpinnings of substance abuse, potentially leading to the improved methods to diagnose those at risk and to help develop better therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Substance abusers
* Allow for blood draw

Exclusion Criteria:

* Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 1992-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Uhl, M.D., Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Noble EP, Blum K, Khalsa ME, Ritchie T, Montgomery A, Wood RC, Fitch RJ, Ozkaragoz T, Sheridan PJ, Anglin MD, et al. Allelic association of the D2 dopamine receptor gene with cocaine dependence. Drug Alcohol Depend. 1993 Oct;33(3):271-85. doi: 10.1016/0376-8716(93)90113-5. PMID 8261891
- [Background] Clark CJ, Downie CC. A method for the rapid determination of the number of patients to include in a controlled clinical trial. Lancet. 1966 Dec 17;2(7477):1357-8. doi: 10.1016/s0140-6736(66)92098-8. No abstract available. PMID 4162809
- [Background] Grandy DK, Litt M, Allen L, Bunzow JR, Marchionni M, Makam H, Reed L, Magenis RE, Civelli O. The human dopamine D2 receptor gene is located on chromosome 11 at q22-q23 and identifies a TaqI RFLP. Am J Hum Genet. 1989 Nov;45(5):778-85. PMID 2573278
- [Background] Hill SY, Armstrong J, Steinhauer SR, Baughman T, Zubin J. Static ataxia as a psychobiological marker for alcoholism. Alcohol Clin Exp Res. 1987 Aug;11(4):345-8. doi: 10.1111/j.1530-0277.1987.tb01323.x. PMID 3307504
- [Background] Shigeta Y, Ishii H, Takagi S, Yoshitake Y, Hirano T, Takata H, Kohno H, Tsuchiya M. HLA antigens as immunogenetic markers of alcoholism and alcoholic liver disease. Pharmacol Biochem Behav. 1980;13 Suppl 1:89-94. doi: 10.1016/s0091-3057(80)80014-1. PMID 7243836
- [Background] Smith SS, O'Hara BF, Persico AM, Gorelick DA, Newlin DB, Vlahov D, Solomon L, Pickens R, Uhl GR. Genetic vulnerability to drug abuse. The D2 dopamine receptor Taq I B1 restriction fragment length polymorphism appears more frequently in polysubstance abusers. Arch Gen Psychiatry. 1992 Sep;49(9):723-7. doi: 10.1001/archpsyc.1992.01820090051009. PMID 1355337
- [Background] Uhl GR, Liu QR, Walther D, Hess J, Naiman D. Polysubstance abuse-vulnerability genes: genome scans for association, using 1,004 subjects and 1,494 single-nucleotide polymorphisms. Am J Hum Genet. 2001 Dec;69(6):1290-300. doi: 10.1086/324467. Epub 2001 Nov 6. PMID 11704927
- [Background] Moolchan ET, Radzius A, Epstein DH, Uhl G, Gorelick DA, Cadet JL, Henningfield JE. The Fagerstrom Test for Nicotine Dependence and the Diagnostic Interview Schedule: do they diagnose the same smokers? Addict Behav. 2002 Jan-Feb;27(1):101-13. doi: 10.1016/s0306-4603(00)00171-4. PMID 11800217
- [Background] Uhl GR, Liu QR, Naiman D. Substance abuse vulnerability loci: converging genome scanning data. Trends Genet. 2002 Aug;18(8):420-5. doi: 10.1016/s0168-9525(02)02719-1. PMID 12142011
- [Background] Stein L, Belluzzi J. Second messengers, natural rewards, and drugs of abuse. Clin Neuropharmacol. 1986;9 Suppl 4:205-7. No abstract available. PMID 3032425
- [Background] Uhl GR, Gold LH, Risch N. Genetic analyses of complex behavioral disorders. Proc Natl Acad Sci U S A. 1997 Apr 1;94(7):2785-6. doi: 10.1073/pnas.94.7.2785. No abstract available. PMID 9096294
- [Background] Uhl GR, Persico AM, Smith SS. Current excitement with D2 dopamine receptor gene alleles in substance abuse. Arch Gen Psychiatry. 1992 Feb;49(2):157-60. doi: 10.1001/archpsyc.1992.01820020068010. No abstract available. PMID 1347991
- [Background] Johnson EO, van den Bree MB, Uhl GR, Pickens RW. Indicators of genetic and environmental influences in drug abusing individuals. Drug Alcohol Depend. 1996 May;41(1):17-23. doi: 10.1016/0376-8716(96)01223-9. PMID 8793306
- [Background] Uhl GR. Molecular genetics of substance abuse vulnerability: a current approach. Neuropsychopharmacology. 1999 Jan;20(1):3-9. doi: 10.1016/S0893-133X(98)00061-X. No abstract available. PMID 9885780
- [Background] Wise RA. Action of drugs of abuse on brain reward systems. Pharmacol Biochem Behav. 1980;13 Suppl 1:213-23. doi: 10.1016/s0091-3057(80)80033-5. No abstract available. PMID 6113601
- [Background] Gelernter J, Moises H, Grandy D, et al. Exclusion of schizophrenia triat from regions of the D2 dopamine receptor and prophobilinogen deaminase genes. In: 28th Annual Meeting, American College of Neurophyschopharmacology, December 13, 1980; Maui, Hawaii, Abstracts p.216.
- [Background] Wyatt RJ, Farouk K, Suddath R, Hitri A. The role of dopamine in cocaine use and abuse. Psychiatric Annals 1988; 18:531-534.